CLINICAL TRIAL: NCT05690854
Title: Cardiovascular Magnetic Resonance in Adults With SysTemic Right Ventricle (STAR): From Pathophysiology to Clinical Application
Brief Title: Cardiovascular Magnetic Resonance in Adults With SysTemic Right Ventricle (STAR)
Acronym: STAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Giulia Pasqualin, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: STAR
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Transposition of Great Arteries
MeSH Terms: conditions — Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: The study will include patients aged ≥ 18 years with the diagnosis of L-TGA and D-TGA, who:
  * are admitted to IRCCS Policlinico San Donato, the Adult Congenital Heart Unit or
  * are scheduled for a Cardiovascular Magnetic Resonance examination in this Institution
- Control: The study will include subjects aged ≥ 18 years who will invited for a Cardiovascular Magnetic Resonance examination in our Institution. This group of control will include n=15 of adult healthy subjects. A further inclusion criteria for the control subjects are age and male proportion comparable to those of the TGA group.

SUMMARY:
The main aim of the study is to explore HFs in SRV, comparing their magnitude and direction with that of subpulmonary RV and systemic LV. As a secondary aim, possible association or correlation will be investigated between SRV energetics and: i) patient functional parameters, e.g., the results from cardiopulmonary exercise test (CPET), ii) patient clinical status, including the occurrence of adverse outcome (a composite of death, hospitalization for heart failure, cardiovascular arrest, sustained arrhythmias).

ELIGIBILITY:
Inclusion Criteria:Case group:

The study will include patients aged ≥ 18 years with the diagnosis of L-TGA and D-TGA, who:

* are admitted to UNICCA, the Adult Congenital Heart Unit or
* are scheduled for a Cardiovascular Magnetic Resonance examination in this Institution

Control group:

The study will include subjects aged ≥ 18 years who will invited for a Cardiovascular Magnetic Resonance examination in our Institution. This group of control will include n=15 of adult healthy subjects. A further inclusion criteria for the control subjects are age and male proportion comparable to those of the TGA group.

Exclusion Criteria:

* (case and control group)

  * Subjects with intrabody ferromagnetic material precluding subject's safety
  * Subjects with non CMR-conditional devices
  * Subjects with claustrophobia or breath-holding precluding an adequate CMR and 4D Flow images quality
  * Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of L-loop transposition of great arteries (L-TGA) and D-loop transposition of great arteries (D-TGA) after atrial switch operation (ASO).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Outcome definition | 5 years
  A composite of death, hospitalizations for heart failure, cardiovascular arrest, sustained arrhythmias (≥30 seconds).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy